CLINICAL TRIAL: NCT01089868
Title: Quantification of Therapy Effects After Microsurgery, Percutaneous Irradiation and Chemotherapy by FET-PET Analysis
Brief Title: Usefulness of Therapy Monitoring by Means of [(18)F]Fluoroethyltyrosine-Positron Emission Tomography (FET-PET) in Glioblastoma Multiforme Patients
Status: Completed | Type: Observational
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: Deutsche Krebshilfe e.V., Bonn (Germany) (Other)
Responsible Party: Principal Investigator, Bogdana Suchorska, PI, Ludwig-Maximilians - University of Munich
Other Study IDs: GGN-ZP9
Record Dates: First submitted 2010-03-17; First posted 2010-03-19 (Estimated); Last update posted 2012-08-07 (Estimated); Status verified 2012-08

CONDITIONS: Glioblastoma Multiforme
Keywords: Glioblastoma multiforme; Microsurgery; Stereotactic biopsy; Radiochemotherapy; Temodar; FET PET; Molecular imaging
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA and RNA samples for MGMT methylation and LOH 1p and 19q status analysis
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group A: Patients who suffer from a suspected GBM and will undergo a microsurgical procedure for diagnosis verification. MRI and Positron Emission Tomography (PET) scans are scheduled prior to microsurgery, post microsurgery and after having completed radiochemotherapy and an additional scan after TMZ chemotherapy.
- Group B: Patients enrolled in Group B suffer from a suspected GBM which cannot be accessed microsurgically either due to a an eloquent location of the tumor, or patient's refusal to undergo surgery. In these patients, diagnosis will be obtained by means of stereotactic surgery. After an initial PET and MRI scan prior to biopsy, patients will be monitored by post radiochemotherapy as well as post 3-months chemotherapy MRI/PET scans.

SUMMARY:
The aim of this study is to establish FET-PET as an additional therapy assessment parameter in patients diagnosed with a glioblastoma multiforme receiving radiochemotherapy and adjuvant chemotherapy after previous resection or biopsy.

ELIGIBILITY:
Inclusion Criteria:

* neuroradiologically suspected Glioblastoma multiforme
* histological verification will be obtained either by microsurgery or by stereotactic biopsy. The neuropathological diagnosis will be verified by a reference neuropathologist
* patients will undergo radiochemotherapy subsequent to surgical procedure
* patients older than 18 years
* Karnofsky Performance Score >=70
* pregnant or nursing female patients will not be included in this study
* safe contraceptive methods during the radiochemotherapy and chemotherapy

Exclusion Criteria:

* patients in whom informed consent cannot be obtained due to organic brain syndrome or insufficient language skills
* patients who cannot lie quiet for a time period of app. two hours during the FET-PEt scan
* medical history of a metastatic brain disease
* patients in whom an MRI scan cannot be performed due to claustrophobia metallic protheses or pacemakers etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have been referred to a neurosurgical department for diagnosis and therapy of a brain tumor
Sampling Method: Non-Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2007-01; Primary Completion 2011-06 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Overall Survival | 46 months

SECONDARY OUTCOMES:
Progression Free Survival | 46 months

CONTACTS AND LOCATIONS:
Overall Officials: Joerg C. Tonn, Prof. Dr., Principal Investigator — Department of Neurosurgery, LMU, Munich
Locations (3):
- Germany (3):
  - Department of Stereotactic Neurosurgery, Freiburg im Breisgau, Baden-Wurttemberg
  - University Hospital Munich, Department of Neurosurgery, Munich, Bavaria
  - University Hospital Bonn, Department of Neurosurgery, Bonn, North Rhine-Westphalia

REFERENCES:
- [Derived] Ingrisch M, Schneider MJ, Norenberg D, Negrao de Figueiredo G, Maier-Hein K, Suchorska B, Schuller U, Albert N, Bruckmann H, Reiser M, Tonn JC, Ertl-Wagner B. Radiomic Analysis Reveals Prognostic Information in T1-Weighted Baseline Magnetic Resonance Imaging in Patients With Glioblastoma. Invest Radiol. 2017 Jun;52(6):360-366. doi: 10.1097/RLI.0000000000000349. PMID 28079702